CLINICAL TRIAL: NCT05174533
Title: Prevalence of Cardiovascular Disorders in Patients Aged 40 and More With Schizophrenia
Acronym: SCHIZO-CV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-011-SCHIZO-CV
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Schizophrenia
Keywords: schizophrenia; cardiovascular disorders; prevalence
MeSH Terms: conditions — Schizophrenia; Cardiovascular Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- with schizophrenia: "with schizophrenia" group : patients aged 40 and more with schizophrenia
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — electrocardiogram

SUMMARY:
Schizophrenia is a psychiatric disorder, affecting 600,000 patients in France. Patients with schizophrenia have life expectancy decrease from 10 to 20 years because of cardiovascular death. Cardiovascular risk factors are numerous: inadequate diet, smoking, alcohol consumption, diabetes, obesity. Primary prevention of cardiovascular risk in patients suffering from schizophrenia is difficult because of understaff in general practitioners and psychiatrists.

DETAILED DESCRIPTION:
The aim of the study is to describe prevalence of cardiovascular disorders in patients aged 40 and more with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* aged of 40 and more
* with schizophrenia
* agreeing to participate in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged of 40 and more with schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-05-12 (Estimated); Study Completion 2022-07-12 (Estimated)

PRIMARY OUTCOMES:
QRS morphology | Day 0
  variation of QRS waves according a standard 12-lead ECG

SECONDARY OUTCOMES:
cardiac rhythm | Day 0
  cardiac rhythm disorder according a standard 12-lead ECG

CONTACTS AND LOCATIONS:
Locations (1):
- Epsmd de l'Aisne, Prémontré, Grand Est, France

IPD SHARING:
Plan to Share IPD: No